CLINICAL TRIAL: NCT00134173
Title: Phase 3, Multi-Center, Double-Blind, Randomized, Parallel Group, Coronary Artery Intravascular Ultrasound Evaluation of the Anti-Atherosclerotic Efficacy, Safety, and Tolerability of Fixed Combination CP-529,414/Atorvastatin, Administered Orally, Once Daily (QD) for 24 Months, Compared With Atorvastatin Alone, in Subjects With Angiographically Documented Coronary Heart Disease.
Brief Title: A Coronary IVUS Study to Compare Torcetrapib/Atorvastatin to Atorvastatin Alone in Subjects With Coronary Heart Disease
Acronym: ILLUSTRATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091005
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-04

CONDITIONS: Coronary Disease; Coronary Arteriosclerosis; Hyperlipidemia
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Hyperlipidemias | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To look at ultrasound images taken in the blood vessels of the heart and to look at various lipids in the blood of people with known coronary heart disease

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* angiographic evidence of coronary atherosclerosis

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid.
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors.
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100
Dates: Start 2003-10; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change coronary artery atheroma volume as measured by intravascular ultrasound.

SECONDARY OUTCOMES:
Changes in levels of lipids and other biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (146):
- United States (127):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Los Altos, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Mountain View, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Stockton, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Brandford, Connecticut
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, Guilford, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Atlantis, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Dunedin, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Safety Harbor, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Blue Island, Illinois
  - Pfizer Investigational Site, Merrionette Park, Illinois
  - Pfizer Investigational Site, Rockford, Illinois
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Goshen, Indiana
  - Pfizer Investigational Site, Hobart, Indiana
  - Pfizer Investigational Site, Merrillville, Indiana
  - Pfizer Investigational Site, Davenport, Iowa
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, West Des Moines, Iowa
  - Pfizer Investigational Site, Shawnee Mission, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Bogalusa, Louisiana
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Lewiston, Maine
  - Pfizer Investigational Site, Portland, Maine
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Salisbury, Maryland
  - Pfizer Investigational Site, Takoma Park, Maryland
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Flint, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, Lapeer, Michigan
  - Pfizer Investigational Site, Petoskey, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Saginaw, Michigan
  - Pfizer Investigational Site, Ypsilanti, Michigan
  - Pfizer Investigational Site, Duluth, Minnesota
  - Pfizer Investigational Site, Maplewood, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Ridgewood, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Carlsbad, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Bay Shore, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Flushing, New York
  - Pfizer Investigational Site, Johnson City, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Oneonta, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Troy, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Eden, North Carolina
  - Pfizer Investigational Site, Greensboro, North Carolina
  - Pfizer Investigational Site, Greenville, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Reidsville, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Bellevue, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Clyde, Ohio
  - Pfizer Investigational Site, Defiance, Ohio
  - Pfizer Investigational Site, Fostoria, Ohio
  - Pfizer Investigational Site, Middleburg Heights, Ohio
  - Pfizer Investigational Site, Orange, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Wauseon, Ohio
  - Pfizer Investigational Site, Westlake, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Florence, Oregon
  - Pfizer Investigational Site, Hillsboro, Oregon
  - Pfizer Investigational Site, Doylestown, Pennsylvania
  - Pfizer Investigational Site, Harrisburg, Pennsylvania
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Lancaster, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Wormleysburg, Pennsylvania
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Chattanooga, Tennessee
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Oak Ridge, Tennessee
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Annandale, Virginia
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Falls Church, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Huntington, West Virginia
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Belgium (3):
  - Pfizer Investigational Site, Aalst
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Genk
- Canada (6):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Victoria, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Torono, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Netherlands (2):
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Rotterdam
- Poland (3):
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Warsaw
- Spain (5):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, L´Hospitalet Del Llobregat, Barcelona
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Vigo, Pontevedra
  - Pfizer Investigational Site, Oviedo, Principality of Asturias

REFERENCES:
- [Derived] Nicholls SJ, Tuzcu EM, Brennan DM, Tardif JC, Nissen SE. Cholesteryl ester transfer protein inhibition, high-density lipoprotein raising, and progression of coronary atherosclerosis: insights from ILLUSTRATE (Investigation of Lipid Level Management Using Coronary Ultrasound to Assess Reduction of Atherosclerosis by CETP Inhibition and HDL Elevation). Circulation. 2008 Dec 9;118(24):2506-14. doi: 10.1161/CIRCULATIONAHA.108.790733. Epub 2008 Nov 24. PMID 19029466
- [Derived] Nissen SE, Tardif JC, Nicholls SJ, Revkin JH, Shear CL, Duggan WT, Ruzyllo W, Bachinsky WB, Lasala GP, Tuzcu EM; ILLUSTRATE Investigators. Effect of torcetrapib on the progression of coronary atherosclerosis. N Engl J Med. 2007 Mar 29;356(13):1304-16. doi: 10.1056/NEJMoa070635. Epub 2007 Mar 26. PMID 17387129
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5091005&StudyName=A+Coronary+IVUS+Study+to+Compare+Torcetrapib%2FAtorvastatin+to+Atorvastatin+Alone+in+Subjects+with+Coronary+Heart+Disease